CLINICAL TRIAL: NCT00134524
Title: A Randomized, Sham-Controlled Clinical Study to Evaluate The Effect of the Magnetic Molecular Energizer (MME) on Diabetic Peripheral Neuropathy
Brief Title: The Effects of the Magnetic Molecular Energizer (MME) on Diabetic Peripheral Neuropathy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Advanced Magnetic Research Institute International (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMRI-DPN-01
Record Dates: First submitted 2005-08-22; First posted 2005-08-25 (Estimated); Last update posted 2007-07-10 (Estimated); Status verified 2007-07

CONDITIONS: Diabetic Neuropathies; Pain; Neuralgia
Keywords: Magnetics; Electromagnetics; Diabetic neuropathy; Pain
MeSH Terms: conditions — Diabetic Neuropathies; Pain; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: MME procedure

SUMMARY:
This study is intended to demonstrate that exposure to a high intensity, DC electromagnetic field, as supplied by the investigational device known as the Molecular Magnetic Energizer (MME), will create a clinically meaningful improvement in pain and nerve dysfunction in the feet of patients with diabetic peripheral neuropathy (DPN).

DETAILED DESCRIPTION:
Diabetic peripheral neuropathy (DPN) affects up to 1/2 of diabetics, both type I and II. It contributes to limb amputation, and can cause painful symptoms which are difficult to treat. Application of a high intensity, DC electromagnetic field, as supplied by the investigational device the Magnetic Molecular Energizer (MME) has shown in a pilot study with participants having DPN in their feet, to have created significant improvement in painful symptoms and improved measures of neurologic function in 7 of 10 participants. This study will enroll participants and evaluate them at baseline with regard to pain levels, nerve function and quality of life. They will then be randomized to receive 120 hr exposure to either active MME procedure, or sham procedure. Following the 120 hrs the participants will then receive the same evaluation for pain level, nerve function and quality of life. These evaluations will be repeated a final time 6 months following. The participants will be blinded to whether they receive the active or sham procedure.

The MME procedure consists of laying on a bed with the feet lying in the space between two large electromagnetic coils which, when activated, produce a DC magnetic field measuring 5000 gauss. The participants will lay on the bed with feet in the magnetic field for 8 to 12 hours a day for 10 to 16 days in succession. Breaks are allowed, and no restraints are required. The procedure may be done at night so that participants may sleep.

Pain assessment will be done by self assessment using rating with the Visual Analogue Scale.

Neurologic function will be assessed with Cutaneous Perception Threshold testing using the Neurometer, a commercially available, FDA approved device.

Quality of life assessment will be by the Neuropathy Specific Quality of Life Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diabetic peripheral neuropathy in feet with associated pain/discomfort.
* Stable and controlled diabetes with hemoglobin A1c level less than 9.0% at entry into the study. Diabetes type I or type II accepted.
* Subjects must be able to read English.

Exclusion Criteria:

* Pacemakers, defibrillators, aneurysm clips, cochlear implants, any metallic particles in eyes or ferromagnetic metal shrapnel, projectile or implant in body.
* Pregnant women
* Concurrent neuropathy not due to diabetes.
* Unstable cardiac disease or uncontrolled blood pressure.
* Renal failure
* Active hepatitis
* History of nerve injury to lower extremities.
* History of spinal surgery or total knee arthroplasty
* Current malignancy
* Alcoholism
* History of stroke
* Seizure disorder
* Current use of long acting narcotic medication
* Skin ulceration or breakdown of the lower extremities
* Peripheral vascular disease sufficient to cause extremity pain at rest.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2005-07; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in neurologic function following procedure
Improvement in DPN related pain following procedure
Subject tolerance to the MME procedure

SECONDARY OUTCOMES:
Neurologic function at 6 month follow-up
Pain level at 6 month follow-up
Quality of Life assessments at baseline, post-procedure and 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wayne R Bonlie, MD, Study Director — AMRI International
Locations (5):
- United States (5):
  - AMRI Arizona, Tucson, Arizona
  - AMRI MI, Sterling Heights, Michigan
  - AMRI NC, Mocksville, North Carolina
  - Amri NW Oh, Toledo, Ohio
  - AMRI WA, Renton, Washington

REFERENCES:
- See also: Study sponsor, AMRI International website homepage — http://www.amri-intl.com